CLINICAL TRIAL: NCT07338630
Title: Phrenic Nerve Sparing of the Interscalene Block Alone Versus Combined With Superior Truncus Block During Shoulder Surgery , Prospective Comparative Randomized Study
Brief Title: Comparison of the Interscalene Block Alone Versus Combined With Superior Truncus Block During Shoulder Surgery in Diaphragmatic Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sherif Salah Ismail, Assistant lecturer of Anesthesia and ICU and Pain Management of Sohag University hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Soh-Med--25-11-5MD
Record Dates: First submitted 2025-12-08; First posted 2026-01-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Diaphragm Issues
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: The patients will be allocated to two groups :
  * Group I (30 patients) : Interscalene block alone, we will inject 20 mL of 0.5 % bupivacaine plus 10 mL of 0.9 % normal saline around brachial plexus in the interscalene site under ultrasonograhy.
  * Group S(30 patients): Interscalene block plus Superior truncus block
    1. We will inject 7 mL of 0.5 % bupivacaine plus 3 mL of 0.9 % normal saline ( Total amount 10 ml) around brachial plexus in the interscalene site under ultrasonograhy.
    2. Also we will inject 13 mL of 0.5 % bupivacaine plus 7 mL of 0.9 % normal saline ( Total amount 20 ml) around Superior trunk of brachial plexus under ultrasonagraphy.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block alone (Active Comparator): Interscalene block alone, we will inject 20 mL of 0.5 % bupivacaine plus 10 mL of 0.9 % normal saline around brachial plexus in the interscalene site under ultrasonograhy.
  Interventions: Other: Regional anesthesia in shoulder surgery
- Interscalene block plus Superior truncus block (Active Comparator): 1. We will inject 7 mL of 0.5 % bupivacaine plus 3 mL of 0.9 % normal saline ( Total amount 10 ml) around brachial plexus in the interscalene site under ultrasonograhy.
  2. Also we will inject 13 mL of 0.5 % bupivacaine plus 7 mL of 0.9 % normal saline ( Total amount 20 ml) around Superior trunk of brachial plexus under ultrasonagraphy.
  Interventions: Other: Regional anesthesia in shoulder surgery

INTERVENTIONS:
Other: Regional anesthesia in shoulder surgery — Comparison of the interscalene block alone versus combined with superior truncus block during shoulder surgery in diaphragmatic function

SUMMARY:
Primarily, This study aims to compare between interscalene block alone versus combined with superior truncus block in producing diaphragmatic paralysis and Secondarily aims to evaluate

1. Effect on the pulmonary function.
2. Duration of the sensory and motor block.
3. Postoperative analgesic consumption.
4. Any complications or side effects during shoulder surgery.

DETAILED DESCRIPTION:
Regional anesthesia is central to modern shoulder surgery because it provides excellent perioperative analgesia, reduces opioid consumption, and facilitates early rehabilitation. The interscalene brachial plexus block (ISB) has long been considered the gold-standard single-shot regional technique for shoulder procedures due to its reliable analgesia and surgical anesthesia. However, ISB commonly causes ipsilateral hemidiaphragmatic paresis (HDP) from unintended phrenic nerve blockade, which can produce clinically important declines in pulmonary function and may be poorly tolerated in patients with limited respiratory reserve.

To minimize phrenic involvement while preserving analgesic effectiveness, more selective approaches have been proposed. The superior trunk block (STB) - performed at the level where C5-C6 fibers form the superior trunk - aims to anesthetize the shoulder innervation more distally and thus reduce spread to the phrenic nerve. A landmark randomized trial and subsequent studies reported that STB provides analgesia comparable to ISB while greatly lowering the incidence of HDP (for example, ISB 71% vs STB 5% in one trial). Systematic reviews and meta-analyses since then have reinforced STB as an effective phrenic-sparing alternative for many shoulder procedures.

Despite encouraging data for STB, the literature is not entirely uniform. Some randomized trials and observational reports have found either reduced anesthetic quality with STB or smaller-than-expected reductions in phrenic involvement, particularly when block technique, local anesthetic volume, or patient anatomy differ. Moreover, combining blocks (for example, ISB with selective superior-trunk targeting or other modifications) has been proposed as a strategy to balance surgical anesthesia and respiratory safety, but comparative prospective data examining the effect of ISB alone versus ISB combined with STB on diaphragmatic function are limited. This uncertainty is important because even partial diaphragmatic paresis can degrade postoperative pulmonary mechanics and increase complications in vulnerable patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I, II physical status.
* Aged between 20 and 65 years.
* Male or female.
* Body Mass index (BMI): 18-30 kg/m3.
* Scheduled for shoulder surgery.

Exclusion Criteria:

* Allergy to local anesthetics.
* Infection at the injection site.
* Coagulation disorders.
* Respiratory diseases ( Acute or Chronic) or Chest trauma.
* Multiple traumatized patients.
* Phrenic nerve injury
* Heart failure, Cardiomyopathy.
* Severe organ dysfunction
* Patient refusal

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between interscalene block alone versus combined with superior truncus block inproducing diaphragmatic paralysis | Assessment of diaphragmatic function by diaphragm excursion (DE) and diaphragm thickening fraction (TF) will be measured both before and 30 minutes post-block.
  Assessment of diaphragmatic function by diaphragm excursion (DE) and diaphragm thickening fraction (TF) will be measured both before and 30 minutes post-block. To measure DE, patients will be placed in a supine position, a convex transducer (3.5 ~ 5 MHz) will be used to scan while the right diaphragm through the hepatic window and the left diaphragm through the splenic window, which located near the anterior-axillary line. The craniocaudal movement of the diaphragm will be documented during deep inspiration using M-mode.
  * Complete diaphragmatic paralysis was defined as a 75% ~ 100% reduction in DE, including the occurrence of paradoxical movement.
  * Partial diaphragmatic paralysis was defined as a 25% ~ 75% reduction in DE.
  * No diaphragmatic paralysis was indicated by a DE reduction of less than 25%. To measure TF, patients will be placed in the same position with the head of the bed at 45°degree

SECONDARY OUTCOMES:
Evaluation of the interscalene block alone versus combined with superior truncus block during shoulder surgery on the pulmonary function | Assessment of pulmonary function by a handheld spirometer to measure forced vital capacity (FVC), forced expiratory volume ( FEV1, FEV2) with patients in an upright-seated position pre-block and 30 minutes post-block as well as 2-hours post-surgery
  Assessment of pulmonary function by a handheld spirometer to measure forced vital capacity (FVC), forced expiratory volume ( FEV1, FEV2) with patients in an upright-seated position pre-block and 30 minutes post-block as well as 2-hours post-surgery. Spirometry will be performed three times, with the best effort recorded.
Duration of the sensory and motor block onset, duration of the interscalene block alone versus combined with superior truncus block during shoulder surgery | Sensory, motor block onset time every minute. Sensory, Motor block duration every hour in 1st 6 hours , every 2 hours in 2nd 6 hours
  Sensory block onset time will be assessed at the time from local anesthetics injection by pinprick test which will be preformed with 22-gauge short beveled needle every minute. Sensory block recovery time will be noted every hour in 1st 6 hours, every 2 hours in 2nd 6 hours till recovery of all pain sensation in all dermatomes performed by pinprick test.
  Motor block onset time will be assessed at the time from local anesthetics injection until complete motor block which will be assessed by absence of voluntary movement on asking the patient to elevate his arm every minute. Motor block recovery time will be noted as the time of return of voluntary movement in the arm every hour in 1st 6 hours, every 2 hours in 2nd 6 hours.
Evaluation of postoperative analgesic consumption | 12 hours
  Pain will be evaluated Postoperative immediately every hour in 1st 6 hours, every 2 hours in 2nd 6 hours by Visual Analogue Scale ( VAS) by instructing the patient to point to the position on the line to indicate how much pain they are currently feeling(10).
  * VAS (zero) indicates no pain.
  * VAS ( 1, 2, 3) indicates mild pain.
  * VAS ( 4, 5, 6) indicates moderate pain.
  * VAS ( 7, 8, 9, 10) : indicates severe pain.
Evaluation of any complications or side effects during shoulder surgery | 24 hours
  Any local or systemic complications or side effects will be recorded every 2 hours post operative for 24 hours such as local anesthetic systemic toxicity (LAST), Horner's syndrome, hypoxia, dyspnea, pneumothorax and post-operative nausea and vomiting (PONV).

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Salah Ismail Assistant lecturer of Anesthesia, Principal Investigator — Assistant lecturer of Anesthesia and ICU and Pain Management of Sohag University hospitals